CLINICAL TRIAL: NCT02684500
Title: Evaluation of Superior Mesenteric Artery Diameter and Flow in Aneurysmal Subarachnoid Hemorrhage Patients Undergoing Hypertensive Therapy for Cerebral Artery Vasospasm
Brief Title: Aneurysmal Subarachnoid Hemorrhage and Superior Mesenteric Artery Flow Study
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500830
Record Dates: First submitted 2016-02-08; First posted 2016-02-18 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Intracranial Aneurysm
Keywords: aSAH
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- aneurysmal subarachnoid hemorrhage: Study measurements of the diameter and doppler flow velocity of the superior mesenteric artery (SMA) using abdominal ultrasound in order to evaluate the potential additional risk of non-occlusive mesenteric ischemia (NOMI) and non occlusive bowel necrosis (NOBN) for a aneurysmal subarachnoid hemorrhage in subjects undergoing hypertensive therapy for cerebral vasospasm in SAH, to justify the withholding of enteral nutrition.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Study measurements of the diameter and doppler flow velocity of the superior mesenteric artery (SMA) for a aneurysmal subarachnoid hemorrhage using abdominal ultrasound.
  Other Names: EDGE Ultrasound System

SUMMARY:
The purpose of this research study is to determine if the diameter and flow of the superior mesenteric artery in patients with aneurysmal subarachnoid hemorrhage undergoing hypertensive therapy for cerebral artery vasospasm are effected enough to justify withholding enteral nutrition.

DETAILED DESCRIPTION:
Study measurements of the diameter and Doppler flow velocity of the superior mesenteric artery (SMA) using abdominal ultrasound in order to evaluate the potential additional risk of non-occlusive mesenteric ischemia (NOMI) and non occlusive bowel necrosis (NOBN) in patients undergoing hypertensive therapy for cerebral vasospasm in Aneurysmal Subarachnoid Hemorrhage (aSAH), to justify the withholding of enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with aSAH

Exclusion Criteria:

* Hemodynamic instability
* Already receiving vasopressor therapy
* Non-aneurysmal SAH
* Intracranial hemorrhage of other cause
* Not anticipated to receive hypertensive therapy with vasoactive medications for cerebral vasospasm from SAH or suspected aSAH
* Unable to visualize SMA using ultrasound
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the neurointensive care unit (NICU).Patients admitted to the neurointensive care unit (NICU) with a diagnosis of aSAH or are diagnosed with aSAH while an inpatient at the NICU at and area hospital.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change between baseline and 21 days of abdominal ultrasound measurement of the diameter in the superior mesenteric artery | Change from baseline up to 21 days
Change between baseline and 21 days of abdominal ultrasound measurement of the doppler flow velocity in the superior mesenteric artery | Change from baseline up to 21 days

SECONDARY OUTCOMES:
Number of participants with non-occlusive mesenteric ischemia (NOMI) | Change from baseline up to 21 days
  Number of participants with non-occlusive mesenteric ischemia (NOMI) undergoing hypertension therapy with vasoactive medications for cerebral arterial vasospasm in aneurysmal subarachnoid hemorrhage (aSAH).
Number of participants with non occlusive bowel necrosis (NOBN) | Change from baseline up to 21 days
  Number of participants with non occlusive bowel necrosis (NOBN) undergoing hypertension therapy with vasoactive medications for cerebral arterial vasospasm in aneurysmal subarachnoid hemorrhage (aSAH).

CONTACTS AND LOCATIONS:
Overall Officials: Peggy White, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No